CLINICAL TRIAL: NCT03281395
Title: Rapid Ventricular Pacing During Cerebral Aneurysm Surgery: a Retrospective Study Concerning the Safety for Heart and Brain
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Joke De Wachter, data manager, University Hospital, Antwerp
Other Study IDs: 17/16/205-2
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Cardiac Pacing, Artificial; Aneurysm, Brain; Arteriovenous Malformations, Cerebral
MeSH Terms: conditions — Intracranial Aneurysm; Intracranial Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral aneurysm surgery with RVP: During surgery patients allocated to this group will undergo RVP. Subjects receive Magnetic Resonance Imaging or Computed Tomography as standard of care, pre-and postoperatively. To screen for rapid ventricular pacing induced micro-infarcts, the contralateral hemisphere(contralateral to the hemisphere operated on) and fossa posterior will be evaluated. Troponin levels are determinated preoperatively and 24 hours postoperatively by blood sample as standard of care. Maximum cTnl level and cTnl level 24 hours will be compared.
  Interventions: Procedure: Rapid ventricular pacing (RVP)
- Craniotomy without RVP: No rapid ventricular pacing is applied during surgery. Subjects receive Magnetic Resonance Imaging or Computed Tomography as standard of care, pre-and postoperatively. To screen for induced micro-infarcts, the contralateral hemisphere(contralateral to the hemisphere operated on) and fossa posterior will be evaluated. Troponin levels are determinated preoperatively and 24 hours postoperatively by blood sample as standard of care. Maximum cTnl level and cTnl level 24 hours will be compared.
  Interventions: Procedure: No rapid ventricular pacing

INTERVENTIONS:
Procedure: Rapid ventricular pacing (RVP) — Rapid ventricular pacing (RVP) is a technique to obtain flow arrest for short period of time during dissection of the aneurysm. RVP results in an adequate fall in blood pressure which presents as an on-off phenomenon. RVP technique facilitates the dissection and manipulation of cerebral aneurysms and arteriovenous malformations and can be lifesaving in the case of an intraoperative bleeding or rupture.
  Groups: Cerebral aneurysm surgery with RVP
Procedure: No rapid ventricular pacing
  Groups: Craniotomy without RVP

SUMMARY:
Rapid ventricular pacing (RVP) is a technique to obtain flow arrest for short periods of time during dissection or rupture of the aneurysm. RVP results in an adequate fall of blood pressure which presents as an on-off phenomenon. It is not clear whether repetitive periods of pacing are harmless for the patient. Silent cardiac and cerebral infarcts may be undetected. The investigator will study the safety of RVP, particularly for the heart and the brain, retrograde by studying troponin levels and magnetic resonance imaging or computed tomography.

DETAILED DESCRIPTION:
Rapid ventricular pacing (RVP) is a technique to obtain flow arrest for short periods of time during dissection or rupture of the aneurysm. RVP results in an adequate fall of blood pressure which presents as an on-off phenomenon. The technique facilitates the dissection and manipulation of cerebral aneurysms and arteriovenous malformations (AVMs) and can be lifesaving in the case of an intraoperative bleeding or rupture. In a former study blood pressure and clinical outcome were used as study parameters. However it is not clear whether repetitive periods of pacing are harmless for the patient. Silent cardiac and cerebral infarcts may be undetected if only clinical outcome is taken as a study parameter. In this retrograde study, the investigators will study the safety of RVP, particularly for the heart and the brain, using magnetic resonance imaging or computed tomography and troponin levels. The purpose of this study is to evaluate the effect of repetitive periods of RVP on the oxygenation of the heart and brain using magnetic resonance imaging and troponin levels both markers for ischemia damage.

ELIGIBILITY:
Inclusion Criteria

* elective cerebral aneurysm clipping surgery
* arteriovenous malformation surgery
* craniotomy
* American Society of Anesthesiologists 1,2 and 3

Exclusion Criteria:

* cardiac abnormalities
* coronary heart disease
* valvular heart disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years, schedulled for elective brain surgery and not responding to any of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2013-01-15 (Actual); Study Completion 2013-07-15 (Actual)

PRIMARY OUTCOMES:
Change of cardiac specific enzyme Troponin (cTnl) from preoperative sample (baseline) | A first blood sample is collected immediately preoperative in the operating room. Postoperative samples are taken at 24 hours up to 60 hours after start surgery
  For detection of myocardial injury, the cardiac specific enzyme Troponin(cTnl)is evaluated pre-and postoperatively

SECONDARY OUTCOMES:
Magnetic resonance imaging or computed tomography | Preoperative and within 1 week post surgery
  Magnetic resonance imaging or computed tomography of the brain pre-and postoperatively is used as standard of care. To screen for RVP induced micro-infarcts, the contralateral hemisphere(contralateral to the hemisphere operated on)and fossa posterior will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD, Principal Investigator — University Hospital, Antwerp; Tomas Menovsky, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium